CLINICAL TRIAL: NCT04882501
Title: Effects of Aromatherapy in Decreasing Nausea Levels in the Post-operative Bariatric Patient Population on a Surgical Unit
Brief Title: Effects of Aromatherapy on Nausea Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U19-07-3670
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Nausea, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Single blinded, parallel arm, placebo- controlled, randomized clinical trial.
Who Masked: Participant
Masking Description: If you agree to participate in the study you will be randomized (assigned by chance) to a product group (product A or product B) and will receive either the active intervention or placebo. There is a 50% or 1 in 2 chance of you receiving either product A or product B upon your initial complaint of nausea when on the Surgical Unit. You will receive a one-time dose for your nausea using either product A or product B based on trial randomization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Actual aromatherapy product (Active Comparator): QUEASEEase quick tab Aromatherapy product 50 % chance of participant receiving based on randomization
  Interventions: Other: QUEASEEase aromatherapy quick tab
- Placebo product (Placebo Comparator): Placebo product (normal saline) 50% chance of participant receiving based on randomization
  Interventions: Other: Placebo product

INTERVENTIONS:
Other: QUEASEEase aromatherapy quick tab — Once patient complains of nausea above intervention will be administered for 5 minutes and nausea level reassessed.
  Arms: Actual aromatherapy product
Other: Placebo product — Once patient complains of nausea above intervention will be administered for 5 minutes and nausea level reassessed.
  Arms: Placebo product

SUMMARY:
Aromatherapy is the therapeutic use of essential oils from plants for the improvement of physical, emotional, and spiritual well-being. Healthcare providers play an important role in improving the care of patients with nausea. Aromatherapy is a complementary therapy that may help with post-operative nausea in the adult post-operative bariatric patient population.

The purpose of this study is to evaluate the effects of aromatherapy intervention on nausea levels with post-operative bariatric patients once they are on the surgical unit.

DETAILED DESCRIPTION:
Subjects will be provided with information about this research study by the following means: a member of the research team- Inova Medical Group (IMG) Nurse Practitioners will discuss the research study during the patient's second pre-operative visit; study information will be uploaded to their MyChart portal; and flyers will be available in the IMG office (refer to appendix A: IMG office flyer). Interested patients will be able to fill out a brief form (refer to appendix B: Interested patient card) requesting to be contacted for further information, this form will be placed in a secure box at the reception desk or the patients can indicate interest by contacting one of the research team members. A member of the research team may need to access medical record information in order to confirm potential patient's phone number and or email address for further contact. A member of the research team will contact any interested patients and answer any questions regarding the research study. Consent will be obtained while the patient is in the peri-operative holding area on day of surgery by a member of the research team, excluding the IMG Nurse Practitioners. The research team member will determine if the patient is eligible for the study, discuss the study, answer any questions, and obtain consent (refer to appendix C: Consent). All members of the research team have completed Informed Consent Training. Once the consented post-operative bariatric patient complains of initial nausea on the Surgical Unit, the direct care nurse or research team member will ask the patient to rate their nausea level using a VAS on a 0-3 scale. Patients will be provided with either product A or B based on randomization scheme calculated by SAS (ver.9.4, Cary, NC). The patient will receive a one-time aromatherapy intervention. Nausea levels will be reassessed 5 minutes after the aromatherapy intervention. If the nausea level does not improve after the study drug intervention an antiemetic medication will be offered (refer to appendix D: Data Collection Form A).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age admitted to the Surgical Unit who are experiencing an initial episode of nausea status post laparoscopic/ robotic sleeve gastrectomy, and/or laparoscopic/robotic Roux-En-Y (RNY) surgery, and/or revisional bariatric surgery; must be able to read and speak English; able to follow directions; bariatric surgeon is part of Inova Medical Group (IMG) and patient is an inpatient.

Exclusion Criteria:

* Patients < 18 years of age; non-English speaking; not able to follow directions; inability to smell (anosmia); allergy to peppermint, spearmint, ginger and/or lavender; receiving bariatric surgery for gastroparesis; pregnant or breastfeeding; vulnerable subjects; receiving complementary therapy (healing touch and/or music therapy) or presently enrolled in another research study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Friesen, PhD, RN, Study Director — IHS
Locations (1):
- Inova Fair Oaks Hospital, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inova Fair Oaks Hospital Started April 19, 2021 Ended August 24, 2022
Period: Overall Study
Arm/Group | Actual Aromatherapy Product | Placebo Product
Started | 55 | 58
Completed | 55 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Actual Aromatherapy Product | Placebo Product | Total
Number analyzed (Participants) | 55 | 58 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 58 | 113
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 38 [20 to 69] | 41 [23 to 59] | 39.3 [20 to 69]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: There were male, female and another category
  Participants
    Male | 2 | 4 | 6
    Female | 52 | 54 | 106
    Decline to answer | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 12 | 17
  Not Hispanic or Latino | 50 | 44 | 94
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 14 | 29
  White | 32 | 29 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 13 | 20
Region of Enrollment [Number; unit: participants]
  United States | 55 | 58 | 113

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Nausea as Measured Visual Analog Scale (VAS) From 0-3
Description: Measured participants self reported nausea level pre ( Baseline) and post intervention VAS 0 - no nausea VAS 1- Mild Nausea VAS 2- Moderate Nausea VAS 3 - Severe nausea
Time Frame: Up to 24 hours post operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Actual Aromatherapy Product | Placebo Product
Number analyzed (Participants) | 55 | 58
Participants
  Baseline: VAS O | 0 | 0
  Baseline: VAS 1 | 13 | 13
  Baseline: VAS 2 | 27 | 25
  Baseline: VAS 3 | 15 | 20
  Post- intervention: VAS O | 16 | 12
  Post- intervention: VAS 1 | 20 | 17
  Post- intervention: VAS 2 | 14 | 17
  Post- intervention: VAS 3 | 5 | 12

2. Secondary Outcome: Total Number of Participants Who Received an Anti-emetic Post Study Intervention.
Description: This the number of patients who received an anti- emetic for nausea after receiving post study intervention.
Time Frame: Up to 24 hours post operatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Actual Aromatherapy Product | Placebo Product
Number analyzed (Participants) | 55 | 58
Participants | 48 | 50

ADVERSE EVENTS:
Time Frame: Collected from time of intervention up to 1.4 days post intervention.
Arm/Group | Actual Aromatherapy Product | Placebo Product
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/58
Other Adverse Events (participants affected / at risk) | 0/55 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT04882501/Prot_SAP_002.pdf